CLINICAL TRIAL: NCT05976841
Title: National Cohort on the Vascular Ehlers-Danlos Syndrome (SEDv)
Brief Title: SEDVasc (RaDiCo Cohort) (RaDiCo-SEDVasc)
Status: Active, not recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C15-65
Record Dates: First submitted 2023-07-18; First posted 2023-08-04 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Ehlers-Danlos Syndrome, Vascular Type
MeSH Terms: conditions — Ehlers-Danlos Syndrome, Type IV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to describe the natural course of vascular Ehlers-Danlos syndrome, in particular the order of appearance of different types of complications (arterial, digestive, pulmonary and uterine).

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this study have to fulfil all of the following criteria:

* Patients (adults and children) with genetically-proven vEDS (presence of a pathogenic mutation at the COL3A1 gene);
* Patients (or his/her legal guardian) who does not oppose to his/her personal data collection.

There are no exclusion criteria for this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed as vEDS on a positive genetic testing on the COL3A1 gene.
Sampling Method: Non-Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Description of the natural course of vascular Ehlers-Danlos syndrome (vEDS) based on anatomical criteria (number and type of arterial lesions or angioscanner or MRI) | Through study completion, an average of 3 years
Description of the natural course of vascular Ehlers-Danlos syndrome (vEDS) based on functional criteria (spontaneous arterial, digestive, obstetrical and pulmonary events) | Through study completion, an average of 3 years
Description of the natural course of vascular Ehlers-Danlos syndrome (vEDS) based on surgical criteria (types and complications) | Through study completion, an average of 3 years
Description of the natural course of vascular Ehlers-Danlos syndrome (vEDS) based on evaluation of the quality of life (impact on daily life, social life and professional activity) | Through study completion, an average of 3 years
Description of the natural course of vascular Ehlers-Danlos syndrome (vEDS) based on evaluation of mortality (death, disability) | Through study completion, an average of 3 years
Description of the natural course of vascular Ehlers-Danlos syndrome (vEDS) based on the presence of complications at delivery or after C-section | Through study completion, an average of 3 years

SECONDARY OUTCOMES:
Study of prospective genotype-phenotype relationships | Through study completion, an average of 3 years
  Mutations of the COL3A1 gene are stratified within 5 classes (Frank et al. Eur J Hum Genet 2015):
  1. Glycine substitutions,
  2. splice-site and in-frame insertions-deletions,
  3. variants leading to haplo-insufficiency,
  4. non-glycine missense variants within the triple helix,
  5. non-glycine missense variants or in-frame insertions-deletions, in the N- or C-terminal part of the protein
  An association study between the type of mutation in the COL3A1 gene (individually or combined in two groups: (a+b) versus (c+d+e)) and the clinical phenotype or co-factors of morbidity (medication, lifestyle, smoking, physical activity…) will be performed. This study will be based on explicative multivariate analysis (e.g.: PCA, Logistic regression, ect.) and relevant association will be quantified by the corresponding correlation coefficient.
Study of the intrafamilial phenotypes relationships | Through study completion, an average of 3 years
  This study will be based on an explicative multivariate analysis (eg: PCA, Logistic regression, ect.) and relevant associations will be quantified by the corresponding correlation coefficients. Distribution of clinical symptoms with a positive correlation with the family history, will be displayed and illustrated by appropriate graphic method (Bar chart, box plot, forest plot, etc.).
Evaluation of the global cost of vEDS cares | Through study completion, an average of 3 years
  The analysis of the global cost of vEDS cares will be detailed by type of expenditure. The average cost will be estimated with health-care payer's perspective, i.e. the French health insurance system.
  After estimating the average global cost of vEDS cares, including both standard pathway's cost and vEDS' cost, a Tornado diagram will analyse the impact of the change of one or more parameters used in the analysis process. This will allow us to identify which parameters have an impact on the result by introducing uncertainties on values used. These parameters will vary in a range obtained by literature review, expert opinion or arbitrarily by simulation on a normal distribution.
  All the results will be drafted in statistical medico-economic analysis report to be presented to all investigators at the end of the study.
Evaluation of the therapeutic management | Through study completion, an average of 3 years
  A descriptive analysis of the different types of medication (celiprolol alone or associated to another drug) and their association to disease progression and life style will be performed by evaluating the number of lesions and/or the increased severity of the lesions and/or the appearance of lesions at different anatomical site.
Assessment of the correlation between the diffusion of arterial lesions and the occurrence of cardiovascular complication | Through study completion, an average of 3 years
Assessment of the repercussions of vEDS on patients' quality of life evaluated through scores of quality of life questionnaire Short-Form Health Survey (SF-36) | Through study completion, an average of 3 years
Assessment of the repercussions of vEDS on patients' quality of life evaluated through scores of quality of life questionnaire Short-Form Health Survey (SF-10) | Through study completion, an average of 3 years
Assessment of the repercussions of vEDS on patients' quality of life evaluated through scores of quality of life questionnaire HADS | Through study completion, an average of 3 years
Assessment of the repercussions of vEDS on patients' quality of life evaluated through scores of quality of life questionnaire socio-professional life | Through study completion, an average of 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Xavier JEUNEMAITRE, Principal Investigator — INSERM UMR S970
Locations (17):
- France (17):
  - Centre Hospitalier Universitaire Angers, Angers
  - Hôpital Saint-André, Bordeaux
  - Hôpital de la Cavale Blanche, Brest
  - Hôpital Côte de Nacre, Caen
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - Hôpital Michallon, Grenoble
  - Hôpital Claude Huriez, Lille
  - Hôpital Edouard Herriot, Lyon
  - Hôpital Femme Mère Enfant, Lyon
  - Hôpital de la Timone, Marseille
  - Hôpital Saint-Eloi, Montpellier
  - Hôpital Brabois, Nancy
  - Hôpital Hôtel Dieu, Nantes
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Nord, Saint-Etienne
  - Hôpital Rangueil, Toulouse
  - Hôpital Trousseau, Tours

IPD SHARING:
Plan to Share IPD: No